CLINICAL TRIAL: NCT01924689
Title: Phase I Safety Study of Intratumoral Injection of Clostridium Novyi-NT Spores in Patients With Treatment-refractory Solid Tumor Malignancies
Brief Title: Safety Study of Intratumoral Injection of Clostridium Novyi-NT Spores to Treat Patients With Solid Tumors That Have Not Responded to Standard Therapies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioMed Valley Discoveries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BVDCNV2
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Solid Tumor Malignancies
Keywords: Phase 1; Metastatic Disease; Solid Tumor; Malignancy; Metastases; Clinical Trial; Hypoxia; Necrosis; Intratumoral; Locally advanced cancer; Immunotherapy; Sarcoma; Chordoma; Bacteriolytic
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Hypoxia; Necrosis; Sarcoma; Chordoma | interventions — Bacterial Load

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clostridium novyi-NT spores (Experimental)
  Interventions: Biological: Clostridium novyi-NT spores

INTERVENTIONS:
Biological: Clostridium novyi-NT spores — Phase 1 study: It will be an escalating dose design, with no intracohort escalation. The first cohort dose will begin at 1 x 10(4) spores/kg and will escalate by tripling through 5 cohorts up to 100 x 10(4) spores/kg.
  Other Names: bacteria; anaerobic bacteria

SUMMARY:
This protocol will examine the safety of intratumoral administration of Clostridium Novyi-NT spores in patients with treatment-refractory solid tumor malignancies. This investigational study will measure anti-tumor activity of C. novyi-NT administered intratumoral in patients with treatment-refractory solid tumor malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of an advanced solid tumor malignancy. There must be a target tumor which is measureable, palpable or clearly identifiable under ultrasound or radiographic guidance and amenable to percutaneous injection of C. novyi-NT spores. The targeted lesion must have a longest diameter ≥ 1 cm and ≤ 12 cm and be measurable as defined by RECIST 1.1 criteria. The target lesion must not be located in either the thoracic, abdominal or pelvic cavities or in the brain. There must be no clinical, no functional, and no radiographic evidence of bone involvement at the site of the target lesion.
2. History of prior treatment with at least one line of systemic anticancer therapy, when an approved systemic therapy is available, and no curative option is available for continued treatment.
3. At least 4 weeks have elapsed since the completion of major surgery, and the patient has fully recovered from this surgery and any post-surgical complications.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less.
5. Patient is at least 18 years of age.
6. Patient is capable of giving informed consent.
7. Patient of childbearing potential (defined by the clinical sites' standards) is using adequate birth control measures (e.g., barrier method with spermicide; intrauterine device; implantable or injectable hormonal contraceptives; surgical sterilization) for the duration of the study and will continue to use such precautions for 12 months after receiving treatment.
8. Patient has no significant valvular heart disease (trace or mild valvular stenosis or regurgitation is allowed).
9. Patient is able to stay within 45 minutes driving time of an emergency room for 28 days after doing.
10. The patient has a caregiver for 28 days after dosing.

Exclusion Criteria:

1. Positive pregnancy test.
2. Serum creatinine level > 1.5 x the upper limit of normal (ULN), chronic renal failure requiring hemodialysis or peritoneal dialysis.
3. Patient has any of the following hematologic parameters:

   * Platelet count equal to or less than 100,000/mm3
   * Hemoglobin less than 9.0 g/dL
   * Absolute neutrophil count (ANC) less than 1,000 /mm3
4. Oxygen saturation (Sp02) of less than 95% on room air.
5. Mean arterial blood pressure (BP) of less than 70 mmHg.
6. Glasgow Coma Score (GCS) of less than 15.
7. Treatment with an investigational drug within the past 30 days or 5 half-lives of that drug, whichever is shorter.
8. Documented primary brain malignancy or brain metastases.
9. Clinically significant ascites or clinical evidence or history of portosystemic hypertension or cirrhosis.
10. Laboratory evidence of hepatic dysfunction indicated by any of the following:

    * Bilirubin ≥ 1.5 x the ULN
    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) above 2.5X the ULN
    * Alkaline phosphatase above 2.5X the ULN
    * International normalized ratio (INR) greater than 1.3
11. Patient has a foreign body which in the opinion of the treating investigator could be difficult to manage in case of infection (e.g. prosthetic hip).
12. Clinically significant pleural effusion.
13. Clinically significant pericardial effusion, circumferential pericardial effusion, or any effusion greater than 1.0 cm at any location around the heart.
14. Need for ongoing treatment with an immunosuppressive agent.
15. History of solid organ transplantation (with the exception of a corneal transplant > 3 months prior to screening).
16. History of an ischemic insult in the previous 12 months (myocardial infarction, cerebral vascular accident, ischemic tissue from injury, transient ischemic attack.
17. History of a significant medical illness deemed by the PI or local investigators as unsuitable for the trial. For example:

    i. Symptomatic congestive heart failure ii. Psychiatric Illness/social situation that may make study dangerous iii. Unstable angina pectoris
18. Asplenia.
19. Antibiotic allergies that would preclude treatment for a C. novyi-NT infection.
20. Treatment with antibiotics within 2 weeks (14 days) of dosing.
21. Active and clinically significant systemic or localized infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - UT M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Janku F, Zhang HH, Pezeshki A, Goel S, Murthy R, Wang-Gillam A, Shepard DR, Helgason T, Masters T, Hong DS, Piha-Paul SA, Karp DD, Klang M, Huang SY, Sakamuri D, Raina A, Torrisi J, Solomon SB, Weissfeld A, Trevino E, DeCrescenzo G, Collins A, Miller M, Salstrom JL, Korn RL, Zhang L, Saha S, Leontovich AA, Tung D, Kreider B, Varterasian M, Khazaie K, Gounder MM. Intratumoral Injection of Clostridium novyi-NT Spores in Patients with Treatment-refractory Advanced Solid Tumors. Clin Cancer Res. 2021 Jan 1;27(1):96-106. doi: 10.1158/1078-0432.CCR-20-2065. Epub 2020 Oct 12. PMID 33046513

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 7 study centers in the United States. A total of 24 patients were enrolled at 4 study centers. Three study centers did not enroll patients.
Pre-assignment Details: Patients who provided informed consent underwent screening procedures within the 21 days preceding C. novyi-NT (Clostridium novyi-Non-Toxic) spore administration. Patients reported to the clinical site 24 hours prior to study Day 0 to reconfirm eligibility and for baseline assessments. Assessments were done as per the schedule of assessment.
Groups:
- Cohort 1: Patients received only single dose of C. novyi-NT spores (Cohort 1: 1 x 10^4 spores) as an intratumoral (IT) injection, per protocol (pp).
- Cohort 2: Patients received only single dose of C. novyi-NT spores (Cohort 2: 3 x 10^4 spores) as an IT injection, pp.
- Cohort 3: Patients received only single dose of C. novyi-NT spores (Cohort 3: 10 x 10^4 spores) as an IT injection, pp.
- Cohort 4: Patients received only single dose of C. novyi-NT spores (Cohort 4: 30 x 10^4 spores) as an IT injection, pp.
- Cohort 5: Patients received only single dose of C. novyi-NT spores (Cohort 5: 100 x 10^4 spores) as an IT injection, pp.
- Cohort 6: Patients received only single dose of C. novyi-NT spores (Cohort 6: 300 x 10^4 spores) as an IT injection, pp.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Started | 3 | 3 | 4 | 6 | 6 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 4 | 6 | 6 | 2
Not completed — Death | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Disease progression | 0 | 0 | 2 | 0 | 3 | 2
Not completed — New therapy or study | 3 | 2 | 1 | 4 | 2 | 0
Not completed — Withdrawal of consent | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Cohort 1: 1 x 10^4 spores
- Cohort 2: Cohort 2: 3 x 10^4 spores
- Cohort 3: Cohort 3: 10 x 10^4 spores
- Cohort 4: Cohort 4: 30 x 10^4 spores
- Cohort 5: Cohort 5: 100 x 10^4 spores
- Cohort 6: Cohort 6: 300 x 10^4 spores
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Total
Number analyzed (Participants) | 3 | 3 | 4 | 6 | 6 | 2 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (14.50) | 55.3 (8.08) | 48.3 (14.13) | 57.2 (12.72) | 59.2 (9.85) | 65.0 (0) | 56.0 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 3 | 2 | 0 | 12
  Male | 1 | 1 | 1 | 3 | 4 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 4 | 6 | 5 | 2 | 22
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 0 | 0 | 2
  White | 2 | 2 | 4 | 6 | 6 | 2 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment-emergent Adverse Events (TEAE)
Description: To determine the safety profile of C. novyi-NT in humans with treatment-refractory solid tumor malignancies when administered as a single IT injection.
  CTCAE: Common Terminology Criteria for Adverse Events
Time Frame: From screening until follow-up visit (up to 12 months)
Population: The safety data set included all patients who received any amount of C. novyi-NT, the investigational medicinal product (IMP). Patients were included in the safety analysis according to the dose of IMP received.
Measure: Number; unit: Patients
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 4 | 6 | 6 | 2
Patients
  All TEAEs | 3 | 3 | 4 | 6 | 6 | 2
  Related TEAEs | 2 | 3 | 2 | 4 | 3 | 2
  CTCAE Grade 1 TEAEs | 3 | 3 | 4 | 5 | 6 | 2
  CTCAE Grade 2 TEAEs | 1 | 3 | 4 | 3 | 2 | 2
  CTCAE Grade 3 TEAEs | 1 | 3 | 2 | 3 | 3 | 2
  Life-Threatening TEAEs | 0 | 1 | 0 | 1 | 0 | 2
  Deaths | 0 | 1 | 0 | 1 | 0 | 0
  Serious TEAEs | 1 | 2 | 1 | 4 | 3 | 2

2. Primary Outcome: Number of Patients With Adverse Events Qualified as Dose Limiting Toxicities (DLTs)
Description: To determine the DLTs of C. novyi-NT in humans with treatment-refractory solid tumor malignancies when administered as a single IT injection.
Time Frame: From screening until follow-up visit (up to 12 months)
Population: The safety data set included all patients who received any amount of C. novyi-NT, IMP. Patients were included in the safety analysis according to the dose of IMP received.
Measure: Number; unit: Patients
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 4 | 6 | 6 | 2
Patients
  Patient with any AEs qualified as DLTs | 0 | 0 | 0 | 1 | 0 | 2
  Patient with Gas gangrene qualified as DLTs | 0 | 0 | 0 | 0 | 0 | 1
  Patient with Sepsis qualified as DLTs | 0 | 0 | 0 | 1 | 0 | 1

3. Secondary Outcome: Percentage Change in Tumor Size From Baseline of the Target Injected Lesion, Measured by Computed Tomography (CT) Scans or Magnetic Resonance Imaging (MRI) Scans
Description: To document preliminary anti-tumor activity of the injected lesion after administering a single IT injection of C. novyi-NT in humans with treatment-refractory solid tumor malignancies. Response and progression was evaluated using the international criteria proposed by the RECIST 1.1. Objective responses were measured by serial CT or MRI scans of the injected lesion and sites of metastatic involvement. Overall response, based on CT/MRI scan results, was based on observation of measurable and non-measurable disease as compared to baseline and nadir in target and non-target tumors per RECIST 1.1.
  Change from baseline is presented.
Time Frame: At screening, at follow up (at 1, 2, 4, and 8 months (±2 days) after dosing)
Population: The efficacy data set or full analysis set consisted of all patients in the safety population who had both a baseline tumor assessment and at least one post-baseline tumor assessment. Patients were included in the analysis according to the dose of IMP received.
Measure: Number; unit: Percentage of change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 4 | 6 | 6 | 2
Percentage of change
  Patient 1, Month 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Patient 1, Month 1 | 1.32 |  |  |  |  |
  Patient 1, Month 2: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Patient 1, Month 2 | -23.68 |  |  |  |  |
  Patient 2, Month 1 and Month 2: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Patient 2, Month 1 and Month 2 | 0 |  |  |  |  |
  Patient 3, Month 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Patient 3, Month 1 | 19.23 |  |  |  |  |
  Patient 4, Month 1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Patient 4, Month 1 |  | -21.90 |  |  |  |
  Patient 4, Month 2: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Patient 4, Month 2 |  | 0 |  |  |  |
  Patient 5, Month 1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Patient 5, Month 1 |  | 11.54 |  |  |  |
  Patient 6, Month 1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Patient 6, Month 1 |  | 10.71 |  |  |  |
  Patient 6, Month 2: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Patient 6, Month 2 |  | 32.14 |  |  |  |
  Patient 7, Month 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Patient 7, Month 1 |  |  | NA — This patient did not have tumor assessments performed at Month 1 |  |  |
  Patient 8, Month 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Patient 8, Month 1 |  |  | -20 |  |  |
  Patient 9, Month 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Patient 9, Month 1 |  |  | -1.85 |  |  |
  Patient 10, Month 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Patient 10, Month 1 |  |  | 6.67 |  |  |
  Patient 11, Month 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Patient 11, Month 1 |  |  |  | -2.22 |  |
  Patient 11, Month 2: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Patient 11, Month 2 |  |  |  | 15.56 |  |
  Patient 12, Month 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Patient 12, Month 1 |  |  |  | 13.56 |  |
  Patient 12, Month 2: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Patient 12, Month 2 |  |  |  | 1.69 |  |
  Patient 12, Month 4: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Patient 12, Month 4 |  |  |  | -13.56 |  |
  Patient 12, Month 8: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Patient 12, Month 8 |  |  |  | 13.56 |  |
  Patient 13, Month 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Patient 13, Month 1 |  |  |  | 26.61 |  |
  Patient 13, Month 2: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Patient 13, Month 2 |  |  |  | 42.20 |  |
  Patient 14, Month 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Patient 14, Month 1 |  |  |  | 14.29 |  |
  Patient 14, Month 2: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Patient 14, Month 2 |  |  |  | 14.29 |  |
  Patient 15, Month 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Patient 15, Month 1 |  |  |  | 16.95 |  |
  Patient 16, Month 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Patient 16, Month 1 |  |  |  | -11.76 |  |
  Patient 16, Month 2: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Patient 16, Month 2 |  |  |  | -14.29 |  |
  Patient 17, Month 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Patient 17, Month 1 |  |  |  |  | -7.14 |
  Patient 17, Month 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Patient 17, Month 2 |  |  |  |  | 0 |
  Patient 17, Month 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Patient 17, Month 4 |  |  |  |  | 3.57 |
  Patient 17, Month 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Patient 17, Month 8 |  |  |  |  | 10.71 |
  Patient 18, Month 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Patient 18, Month 1 |  |  |  |  | 30.23 |
  Patient 18, Month 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Patient 18, Month 2 |  |  |  |  | 86.05 |
  Patient 19, Month 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Patient 19, Month 1 |  |  |  |  | -6.67 |
  Patient 19, Month 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Patient 19, Month 2 |  |  |  |  | 6.67 |
  Patient 20, Month 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Patient 20, Month 1 |  |  |  |  |  | 48.24
  Patient 20, Month 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Patient 20, Month 2 |  |  |  |  |  | 23.53
  Patient 21, Month 1, Month 2, Month 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Patient 21, Month 1, Month 2, Month 4 |  |  |  |  |  | NA — This patient did not have tumor assessments performed at Month 1
  Patient 22, Month 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Patient 22, Month 1 |  |  |  |  | 12.20 |
  Patient 22, Month 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Patient 22, Month 2 |  |  |  |  | 19.51 |
  Patient 23, Month 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Patient 23, Month 1 |  |  |  |  | 3.13 |
  Patient 23, Month 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Patient 23, Month 2 |  |  |  |  | 18.75 |
  Patient 24, Month 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Patient 24, Month 1 |  |  |  |  | 19.30 |

4. Secondary Outcome: Number of Patients With RECIST Assessment on the Injected Lesion
Description: To document preliminary anti-tumor activity of the injected lesion after administering a single IT injection of C. novyi-NT in humans with treatment-refractory solid tumor malignancies. The evaluation of anti-tumor activity included a response for the injected lesion.
  Response and progression was evaluated using the international criteria proposed by the RECIST 1.1. Objective responses were measured by serial CT or MRI scans of the injected lesion and sites of metastatic involvement. Overall response, based on CT/MRI scan results, was based on observation of measurable and non-measurable disease as compared to baseline and nadir in target and non-target tumors per RECIST 1.1.
Time Frame: At follow up (at 1 and 2, 4, and 8 months (±2 days) after dosing)
Population: as for outcome 3
Measure: Number; unit: Patients
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 4 | 6 | 6 | 2
Patients
  Month 1, Complete Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 1, Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 1, Partial Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 1, Partial Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 1, Stable Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 1, Stable Disease | 3 | 3 | 3 | 6 | 6 | 0
  Month 1, Progressive Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 1, Progressive Disease | 0 | 0 | 0 | 0 | 0 | 1
  Month 1, Unknown: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 1, Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Month 2, Complete Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 2, Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 2, Partial Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 2, Partial Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 2, Stable Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 2, Stable Disease | 2 | 0 | 0 | 4 | 3 | 0
  Month 2, Progressive Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 2, Progressive Disease | 0 | 2 | 0 | 1 | 2 | 1
  Month 2, Unknown: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 2, Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Month 4, Complete Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 4, Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 4, Partial Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 4, Partial Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 4, Stable Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 4, Stable Disease | 0 | 0 | 0 | 1 | 1 | 0
  Month 4, Progressive Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 4, Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0
  Month 4, Unknown: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 4, Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Month 8, Complete Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 8, Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 8, Partial Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 8, Partial Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 8, Stable Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 8, Stable Disease | 0 | 0 | 0 | 0 | 0 | 0
  Month 8, Progressive Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 8, Progressive Disease | 0 | 0 | 0 | 1 | 1 | 0
  Month 8, Unknown: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 8, Unknown | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Patients With Overall RECIST Response
Description: To document preliminary anti-tumor activity of an overall response after administering a single IT injection of C. novyi-NT in humans with treatment-refractory solid tumor malignancies. The evaluation of anti-tumor activity included an overall response.
Time Frame: At follow up (at 1 and 2, 4, and 8 months (±2 days) after dosing)
Population: as for outcome 3
Measure: Number; unit: Patients
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 4 | 6 | 6 | 2
Patients
  Month 1, Complete Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 1, Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 1, Partial Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 1, Partial Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 1, Stable Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 1, Stable Disease | 2 | 2 | 3 | 6 | 6 | 0
  Month 1, Progressive Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 1, Progressive Disease | 1 | 1 | 0 | 0 | 0 | 0
  Month 1, Unknown: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 1, Unknown | 0 | 0 | 0 | 0 | 0 | 1
  Month 2, Complete Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 2, Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 2, Partial Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 2, Partial Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 2, Stable Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 2, Stable Disease | 2 | 0 | 0 | 4 | 3 | 0
  Month 2, Progressive Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 2, Progressive Disease | 0 | 2 | 0 | 1 | 2 | 1
  Month 2, Unknown: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 2, Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Month 4, Complete Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 4, Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 4, Partial Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 4, Partial Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 4, Stable Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 4, Stable Disease | 0 | 0 | 0 | 1 | 1 | 0
  Month 4, Progressive Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 4, Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0
  Month 4, Unknown: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 4, Unknown | 0 | 0 | 0 | 0 | 0 | 0
  Month 8, Complete Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 8, Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 8, Partial Response: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 8, Partial Response | 0 | 0 | 0 | 0 | 0 | 0
  Month 8, Stable Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 8, Stable Disease | 0 | 0 | 0 | 0 | 0 | 0
  Month 8, Progressive Disease: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 8, Progressive Disease | 0 | 0 | 0 | 1 | 1 | 0
  Month 8, Unknown: number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 1
  Month 8, Unknown | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Positive Blood Cultures-Number of Patients With Presence of C. Novyi-NT
Description: To study the presence of circulating C. novyi-NT spores after administration as a single IT injection to humans with treatment-refractory solid tumor malignancies.
Time Frame: At Screening, at Days -1 to 0, at Days 1, 2, 3, 4, 5, 7, at follow up (at 2 months (±2 days) after dosing)
Population: The safety data set included all patients who received any amount of C. novyi-NT, the IMP. Patients were included in the safety analysis according to the dose of IMP received.
  Note: Two patients had positive C.novyi culture at Screening due to contamination, and one patient in Cohort 4 had positive C. novyi culture on Day 3 due to contamination.
Measure: Number; unit: Patients
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 4 | 6 | 6 | 2
Patients
  Scheduled, Screening | 0 | 1 | 0 | 0 | 0 | 1
  Scheduled, Day -1 to Day 0 | 0 | 0 | 0 | 0 | 1 | 0
  Scheduled, Day 1 | 0 | 0 | 0 | 0 | 1 | 1
  Scheduled, Day 2 | 0 | 0 | 0 | 1 | 0 | 0
  Scheduled, Day 3 | 1 | 0 | 0 | 1 | 0 | 0
  Scheduled, Day 4 | 1 | 0 | 0 | 0 | 0 | 0
  Scheduled, Day 5 | 1 | 0 | 0 | 0 | 0 | 0
  Scheduled, Day 7 | 0 | 0 | 0 | 0 | 0 | 1
  Scheduled, Month 2 | 1 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Patients With Cytokine Responses Analyzed
Description: The host immune and inflammatory response to C. novyi-NT spores was measured in routine blood sampling over the course of the study.
  The following table presents the data for the patients who had analyzable cytokine data.
  This table was included to simply indicate the number of patients who participated in the cytokine response analysis.
Time Frame: 2 years
Population: as for outcome 3
Measure: Number; unit: Patients
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 4 | 6 | 6 | 2
Patients | 3 | 3 | 4 | 6 | 6 | 2

8. Secondary Outcome: Number of Patients With Systemic Tumor Antigen Specific T-cell Responses
Description: The host immune and inflammatory response to C. novyi-NT spores was measured in routine blood sampling over the course of the study. Release of T-cell cytokines and effector molecules (interferon [IFN]-γ , Granzyme B, and tumor necrosis factor [TNF]-α) from the patient's own peripheral blood mononuclear cells (PBMCs) treated with allogenic tumor cell line lysates were quantified by Enzyme-Linked Immunosorbent Spot (ELISPOT) assays. A positive response was defined as a frequency that is significantly (p <0.05, two-tailed t-test) greater than the mean of control no-antigen wells and detectable (i.e., >1:100,000).
  No patients were analyzed for Cohort 1 and Cohort 2 based on the original study protocol.
Time Frame: 2 years
Population: as for outcome 3
Measure: Number; unit: Patients
Arm/Group | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 4 | 4 | 1
Patients | 1 | 2 | 3 | 1

9. Secondary Outcome: Number of Patients With Local Tumor-specific T-cell Responses
Description: The host immune and inflammatory response to C. novyi-NT spores was measured in routine blood sampling over the course of the study. Immunostaining for tumor infiltrating cells was analyzed independently by 2 investigators. Respective counting of 3 slides per patient between 5 to 20 fields of vision at 200x were scored using the modified ALLRED scoring method. Respective counts were averaged in each case. Pre and post treatment needle biopsies from injected and non-injected tumors were stained for the presence of tumor infiltrating immune cells.
  No patients were analyzed for Cohort 1 and Cohort 2 based on the original study protocol.
Time Frame: 2 years
Population: as for outcome 3
Measure: Number; unit: Patients
Arm/Group | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 1 | 3 | 3 | 2
Patients | 0 | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: From screening until follow-up visit (up to 12 months)
Description: An Adverse Event (AE) was any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation subject administered an investigational medicinal product, even if it did not have a causal relationship with that product. Any unfavorable or unintended sign, symptom, or disease temporally associated with the use of the study agent, whether or not it was considered study agent-related was considered an AE.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 0/4 | 1/6 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 1/4 | 4/6 | 3/6 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 6/6 | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=4) | Cohort 4 (N=6) | Cohort 5 (N=6) | Cohort 6 (N=2)
Disease progression (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0
Oedema peripheral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gas gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Phantom pain (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Genital swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Limb salvage therapy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Osteosynthesis (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=4) | Cohort 4 (N=6) | Cohort 5 (N=6) | Cohort 6 (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 3 | 2 | 2 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 4 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 4 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 1 | 2 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 1 | 3 | 3 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains confidential information of BioMed Valley Discoveries, Inc. Do not copy or distribute without written permission from the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2014-09-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT01924689/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT01924689/SAP_001.pdf